CLINICAL TRIAL: NCT02362880
Title: Study of Genetic Alzheimer's Disease Mutation Carriers in Preclinical Stages of the Disease: 18F-Florbetaben Positron Emission Tomography Study
Brief Title: Study of Genetic Alzheimer's Disease Mutation Carriers in Preclinical Stages of the Disease 18F-Florbetaben Positron Emission Tomography Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: On 15 January 2019, the sponsor decided to stop the study prematurely due to lack of patient recruitment because of supply problems with 18 F-Florbetaben.
Sponsor: Judit Pich Martínez (Other)
Responsible Party: Sponsor-Investigator, Judit Pich Martínez, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FBB-FAD-2014
Record Dates: First submitted 2015-02-09; First posted 2015-02-13 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mutation carrier (Active Comparator)
  Interventions: Radiation: Florbetaben
- mutation non-carrier (Sham Comparator)
  Interventions: Radiation: Florbetaben

INTERVENTIONS:
Radiation: Florbetaben — single dose of Florbetaben followed by PET scan

SUMMARY:
The main purpose of the study is to assess safety of a single dose of FBB followed by PET scan in individuals at risk of genetic Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult children (> 18 yo) of genetic Alzheimer?s disease patients with a known mutation in PSEN1, APP o PSEN2 genes and who are either cognitively normal (CDR=0) or have mild symptoms of cognitive decline (CDR 0.5 or 1)
* According to the principal investigator, participants must be committed to participate and complete all study procedures.
* Has signed the Informed Consent Form voluntarily to participate in the study

Exclusion Criteria:

* Subjects that are not able to complete the study.
* Any major disease or history of a major disease, especially hepatobilliar disease (AST /ALT ? 5 x ULN) or advanced renal insufficiency (creatinine ? 2 x ULN)
* Current or previous history of alcohol abuse or epilepsy
* Allergic to Florbetaben or any of its constituents
* Multiple drug allergies and/or previous history of contrast allergy.
* Pregnancy or breast feeding or planned pregnancy during the study period
* Any disease or history of disease which, in the opinion of the investigator, can cause disturbance of brain function (e.g. vitamin B12 or folic acid deficiency, disturbed thyroid function)
* Evidence for any other neurological or psychiatric disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse events of a single dose of FBB followed by PET scan in individuals at risk of genetic Alzheimer?s disease. | At baseline, when FBB-PET is performed.
Proportion of FAD mutation carriers that present positive uptake after FBB-PET through visual examination | At baseline, when FBB-PET is performed.

SECONDARY OUTCOMES:
Proportion of FAD mutation carriers presenting standardized uptake value ratios (SUVRs) of FBB-PET higher than 1,4. | baseline
Areas of significant difference (p<0,05) in regional SUVR between FAD mutation carriers and non-carriers. | baseline
Earliest age of positive FBB-PET in FAD mutation carriers. | baseline
Individual cortical areas with positive amyloid deposition at visual or semi-quantitative assessment | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Sánchez, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain